CLINICAL TRIAL: NCT02481622
Title: Inhibition by the Antibody, First Event of Infection by HIV-1 of Uterine Vaginal Tissue
Brief Title: First Event of Infection by HIV-1 of Uterine Vaginal Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6197
Record Dates: First submitted 2015-06-07; First posted 2015-06-25 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2015-11

CONDITIONS: HIV Infection of the Uterine Vaginal Tissues
Keywords: HIV infection; vaginal tissues; uterine tissues
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study aims to characterize the cells infected with HIV over time in different types of vagino-uterine tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age ≤50 years and ≥18 years
* Patients for which surgery like laparoscopy or hysterectomy is necessary as part of a benign pathology.

Exclusion Criteria:

* Patients under 18 years

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women whose age ≤50 years and ≥18 years, for which surgery type laparoscopy or hysterectomy is necessary as part of a benign pathology.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
identification of the first HIV-infected cells by a histological analysis | after surgery, up to 3 weks

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine OHL, MD, Principal Investigator — University Hospital, Strasbourg, France; Christiane OHL, PhD, Study Director — UNISTRA
Locations (1):
- INSERM U1109 - Institut de Virologie 3, rue Koeberlé - 67000 Strasbourg, Strasbourg, France